CLINICAL TRIAL: NCT06352879
Title: Prevalence, Types and Risk Factors of Urinary Incontinence Among Women Attending Primary Healthcare Centers in Baghdad, Iraq.
Brief Title: Prevalence, Types and Risk Factors of Urinary Incontinence Among Women in Baghdad, Iraq.
Status: Recruiting | Type: Observational
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 18-Al-KindyCM
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Urinary Incontinence; Urge Incontinence; Stress Incontinence
Keywords: Urinary Incontinence; Urge incontinence; Stress incontinence; Mixed incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to observe and describe the prevalence, types, and risk factors of urinary incontinence (UI) in adult women attending primary healthcare centers in Baghdad, Iraq. The main questions it aims to answer are:

* What is the prevalence of incontinence among the targeted group?
* What are the types of incontinence and what is the frequency of each type among the targeted group?
* What is the effect of several risk factors on the occurrence and severity of urinary incontinence (including age, job, sexual activity, chronic constipation, chronic cough, parity, largest birth weight, and body mass index)? Participants will be asked to fill out a questionnaire consisting of the Arabic International Consultation On Incontinence Questionnaire-Urinary Incontinence Short Form (Arabic ICIQ-UI SF) in addition to questions about the aforementioned risk factors.

ELIGIBILITY:
Inclusion Criteria:

* women
* Attending the primary healthcare centers in Baghdad, Iraq
* older than 18 years

Exclusion Criteria:

* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women attending primary healthcare centers in Baghdad, Iraq
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Arabic International Consultation On Incontinence Questionnaire-Urinary Incontinence Short Form (Arabic ICIQ-UI SF) | 3 months
  Arabic International Consultation On Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) consists of three-scored items designed to evaluate the frequency of urine leaks (score 0-5), the amount of leaked urine (score 0-6), and the effect urine leakage on the quality of life of the participant (score 0-10). In addition, an unscored item to evaluate the sensed causes of leakage. The scores of the scored items are added together to provide a total score, which ranges from zero to 21. The higher the score, the more severe the urine leakage.

SECONDARY OUTCOMES:
Risk factors for urinary incontinence | 3 months
  the study aim to study the effect of several risk factors on the occurrence and severity of urinary incontinence (including age, job, sexual activity, chronic constipation, chronic cough, parity, largest birth weight, and body mass index).

CONTACTS AND LOCATIONS:
Overall Officials: Harth Mohamed Kamber, FICMS (Uro.), Study Chair — University of Baghdad / Alkindy collage of medicine
Locations (2):
- Iraq (2):
  - Baghdad Al- Karkh Health Directorate, Baghdad
  - Baghdad Al-Russafa Health Directorate, Baghdad